CLINICAL TRIAL: NCT06143852
Title: Comparing Change in Social Media Use and Well-being Among College Students Receiving a One-week Exercise or Mindfulness Intervention
Brief Title: Change in Social Media Use and Well-being Among College Students Receiving a One-week Exercise or Mindfulness Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00025926
Record Dates: First submitted 2023-11-14; First posted 2023-11-22 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Social Media Addiction; Depression, Anxiety; Well-Being, Psychological
MeSH Terms: conditions — Internet Addiction Disorder; Depression; Anxiety Disorders; Psychological Well-Being | interventions — Mindfulness; Exercise

STUDY DESIGN:
Intervention Model Description: Three groups of 1) no intervention, 2) mindfulness, or 3) social media reduction + exercise replacement intervention arms
Masking Description: Both participants and investigators will know which intervention group each participant has been randomized into.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants will not receive an intervention. They will receive instructions to use their social media use as usual.
- Mindfulness (Experimental): Approximately 12-minute mindfulness-style meditations will be completed daily for one week through the Calm platform. Participants can listen to the exercise on the web-enabled version of Calm, or through the smartphone app. The course is entitled "7 Days of Gratitude" and centers around noticing and appreciating things in daily life.
  Interventions: Behavioral: Mindfulness
- Social Media Reduction + Exercise (Experimental): Participants will reduce their social media use by at least 30 minutes daily for one week. Simultaneously, participants will exercise at least 30 minutes daily. Participants are given examples of common exercises (walking, yoga, strength training, etc.), but they are allowed to choose any type, although they are dissuaded from activities with high potential for injury.
  Interventions: Behavioral: Social Media Reduction + Exercise

INTERVENTIONS:
Behavioral: Mindfulness — 12 minute daily guided meditation
  Arms: Mindfulness
Behavioral: Social Media Reduction + Exercise — Reduce social media use at least 30 minutes daily and exercise instead
  Arms: Social Media Reduction + Exercise

SUMMARY:
The investigators will be randomizing 150 college student participants with high levels of social media use into either a 1) control condition (no intervention), a 2) mindfulness meditation cognitive intervention, or 3) a social media reduction + exercise replacement intervention. Participants complete intervention activities daily for one week. The investigators will collect self-report and behavioral measures of social media use and related psychological constructs at three time points: baseline, immediately after the intervention period, and one-week after the intervention period.

DETAILED DESCRIPTION:
The objective of this study is to test two cognitive and behavioral interventions designed to reduce social media use and psychological constructs related to social media use in a sample of university students.

The first cognitive intervention is a mindfulness meditation exercise taken from the Calm app centering around gratitude. Each meditation takes approximately 12 minutes to complete and is to be done daily for one week. The second behavioral intervention is asking participants to reduce social media use for 30 minutes daily for one week and replacing that time with physical exercise of the participants' choosing.

Aim 1: Compare psychological constructs related to mental health (well-being, stress, depression, anxiety, loneliness, social comparisons, etc.) before and after conducting two social media use interventions over a period of one week, compared to a control condition (no intervention).

Aim 2: Compare self-reported and behavioral (smartphone screen shots of social media use screen time) measures of social media use before and after two social media use interventions over a period of over one week, compared to a control condition (no intervention).

Aim 3: Examine mental health and social media use one week after the intervention period is complete (follow up), examining or testing whether effects last beyond the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* The participant is 18 or older.
* The participant must be a Johns Hopkins University student.
* Owning an iPhone or Android smartphone, with frequent use of social media use daily (> 1 hour)
* Enabling and sharing screenshots of your smartphone use metrics, including number of last-week pickups, notifications received, and average screen time.
* Providing consent to participate.
* Only exercising 1 hour or less daily, on average.

Exclusion Criteria:

* younger than 18
* Not a Johns Hopkins University Student
* Doesn't own a smart phone
* Uses smartphone less than 1 hour daily
* Exercises more than 1 hour daily

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Change in Depression, Anxiety and Stress Scale - 21 (DASS-21) | baseline, immediately post intervention, post intervention up to one week
  Score range = 0-63, higher score = worse outcome
Change in World Health Organization Quality of Life (WHOQoL-BREF) scale | baseline, immediately post intervention, post intervention up to one week
  Score range = 13-65, lower score = worse outcome
Change in Smartphone screen time (minutes) for social media use | baseline, immediately post intervention, post intervention up to one week
  Past-week amount of screen time for social media use
Change in Number of Social media use smartphone pick-ups | baseline, immediately post intervention, post intervention up to one week
  Past-week total number of smartphone pick-ups for social media use applications
Change in Percent of time using social media | baseline, immediately post intervention, post intervention up to one week
  Past-week percent of time using social media compared to other smartphone application categories.
Change in Social media use notifications received | baseline, immediately post intervention, post intervention up to one week
  Past-week total number of notifications received for social media use applications

SECONDARY OUTCOMES:
Change in University of California, Los Angeles 3-Item Loneliness Scale | baseline, immediately post intervention, post intervention up to one week
  Score range = 3-9, higher score = worse outcome
Change in The Gratitude Questionnaire, 6-item form (GQ-6) scale | baseline, immediately post intervention, post intervention up to one week
  Score range = 6-42, lower score = worse outcome
Change in Motivations for Electronic Interaction Scale (MEIS) | baseline, immediately post intervention, post intervention up to one week
  Score range = 10-50, higher score = worse outcome
Change in Comprehensive Assessment of Acceptance and Commitment Therapy Processes (CompACT-15) scale | baseline, immediately post intervention, post intervention up to one week
  Score range = 0-138, lower scores = worse outcome
Change in Bergen Social Media Addiction Scale (BSMAS) | baseline, immediately post intervention, post intervention up to one week
  Score range = 6-35, higher score = worse outcome
Change in Fear of Missing Out Scale | baseline, immediately post intervention, post intervention up to one week
  Score range = 10-50, higher score = worse outcome
Change in Hours spent socializing in-person with peers | baseline, immediately post intervention, post intervention up to one week
  Score range = 0-20+ hours of in-person socialization, lower scores = worse outcomes
Change in Number of evenings of past-week recreation | baseline, immediately post intervention, post intervention up to one week
  Score range = 0-7 evenings of recreation, lower scores = worse outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Thrul, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We will discuss as a team the how to share individual participant data with other researchers in a confidential manner.

REFERENCES:
- [Background] Hanley SM, Watt SE, Coventry W. Taking a break: The effect of taking a vacation from Facebook and Instagram on subjective well-being. PLoS One. 2019 Jun 6;14(6):e0217743. doi: 10.1371/journal.pone.0217743. eCollection 2019. PMID 31170206
- [Background] Hou, Y., Xiong, D., Jiang, T., Song, L., & Wang, Q. (2019). Social media addiction: Its impact, mediation, and intervention. Cyberpsychology: Journal of Psychosocial Research on Cyberspace, 13(1), article 4.
- [Background] Hunt, M. G., Marx, R., Lipson, C., & Young, J. (2018). No more FOMO: Limiting social media decreases loneliness and depression. Journal of Social and Clinical Psychology, 37(10), 751-768.
- [Background] Lambert J, Barnstable G, Minter E, Cooper J, McEwan D. Taking a One-Week Break from Social Media Improves Well-Being, Depression, and Anxiety: A Randomized Controlled Trial. Cyberpsychol Behav Soc Netw. 2022 May;25(5):287-293. doi: 10.1089/cyber.2021.0324. Epub 2022 May 3. PMID 35512731
- [Background] Roberts TA, Daniels EA, Weaver JM, Zanovitch LS. "Intermission!" A short-term social media fast reduces self-objectification among pre-teen and teen dancers. Body Image. 2022 Dec;43:125-133. doi: 10.1016/j.bodyim.2022.08.015. Epub 2022 Sep 21. PMID 36152479
- [Background] van Wezel MMC, Abrahamse EL, Vanden Abeele MMP. Does a 7-day restriction on the use of social media improve cognitive functioning and emotional well-being? Results from a randomized controlled trial. Addict Behav Rep. 2021 Jun 15;14:100365. doi: 10.1016/j.abrep.2021.100365. eCollection 2021 Dec. PMID 34938826
- [Background] Vanman EJ, Baker R, Tobin SJ. The burden of online friends: the effects of giving up Facebook on stress and well-being. J Soc Psychol. 2018;158(4):496-507. doi: 10.1080/00224545.2018.1453467. Epub 2018 Apr 9. PMID 29558267
- [Background] Nicuță, E.G., Constantin, T. Take Nothing for Granted: Downward Social Comparison and Counterfactual Thinking Increase Adolescents' State Gratitude for the Little Things in Life. J Happiness Stud 22, 3543-3570 (2021). https://doi.org/10.1007/s10902-021-00382-5.
- [Result] Hall, J.A., Xing, C., Ross. E.M., Johnson, R.M. Experimentally manipulating social media abstinence: results of a four-week diary study. Media Psychology, 2019; 24, 259 - 275